CLINICAL TRIAL: NCT04040491
Title: Single-arm, Multi-center Clinical Study of PD-1 Antibody, Chidamide, Lenalidomide and Gemcitabine for Peripheral T-cell Lymphoma
Brief Title: PD-1 Antibody, Chidamide, Lenalidomide and Gemcitabine for Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20190702
Record Dates: First submitted 2019-07-02; First posted 2019-07-31 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: PD-1; chidamide; lenalidomide; gemcitabine; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Lenalidomide; Gemcitabine

STUDY DESIGN:
Intervention Model Description: 50 patients for newly diagnosed group and 50 patients for relapse/refractory group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Newly diagnosed PTCL (Experimental): PD-1 Antibody: 200mg, d1, Chidamide: 30mg, twice a week, Lenalidomide: 10mg, d1-10 gemcitabine:600mg/m2, d1 and 21 days made one treatment cycle.
  Interventions: Drug: PD-1 blocking antibody, chidamide, lenalidomide and gemcitabine
- Relapse/refractory PTCL (Other): PD-1 Antibody: 200mg, d1, Chidamide: 30mg, twice a week, Lenalidomide: 10mg, d1-10 gemcitabine:600mg/m2, d1 and 21 days made one treatment cycle.
  Interventions: Drug: PD-1 blocking antibody, chidamide, lenalidomide and gemcitabine

INTERVENTIONS:
Drug: PD-1 blocking antibody, chidamide, lenalidomide and gemcitabine — PD-1 blocking antibody inhibits PD-1. Chidamide is an histone deacetylase inhibitor. Lenalidomide is a potent inhibitor of TNF-α. Gemcitabine is a cytosine nucleoside derivative, its main metabolite incorporates into DNA in cells and mainly acts on G1 / S phase.

SUMMARY:
To observe the safety, tolerability and clinical effects of PD-1, chidamide, lenalidomide and gemcitabine in the treatment of newly diagnosed and relapse/refractory peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Patients with peripheral T-cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully with the conventional CHOP regimen. The investigators have been proceeding this trial to evaluate the efficacy and safety of the PD-1, chidamide, lenalidomide and gemcitabine in the treatment of newly diagnosed and relapse/refractory peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* age:14-65 years;Eastern Cooperative Oncology Group (ECOG)score≤3;expected survival≥3 months
* patients with Peripheral T-cell Lymphoma diagnosed by immuno-histochemistry (IHC);
* acceptable hematological indicators, no chemotherapy contraindications;
* total bilirubin ≤ 1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 2.5 x upper age limit (ULN), if the abnormal laboratory parameters are considered to be caused by lymphoma, patients Eligible conditions should be adjusted to be incorporated into the group;
* At least one measurable lesion by CT or PET-CT（Positron Emission Tomography-Computed Tomography）;
* exclude other major diseases, normal heart and lung function;
* Female patients of childbearing age are negative for pregnancy test;
* Cooperate with follow-up;
* There are no other related treatments including traditional Chinese medicine, immunotherapy, and biologic therapy (except for the treatment of anti-bone metastases and other symptoms);
* Signing informed consent *: Pathological histology must be consulted by a pathologist at a provincial hospital.

Exclusion Criteria:

* Patients with ALK-positive Anaplastic Large Cell Lymphoma or angioimmunoblastic T-cell lymphoma
* rejecting providing blood preparation;
* allergic to drug in this study and with metabolic block;
* rejecting adopting reliable contraceptive method in pregnancy or lactation period;
* uncontrolled internal medicine disease(including uncontrolled diabetes,severe incompetence cardiac, lung, liver and pancreas）；
* with severe infection;
* with primary or secondary central nervous system tumor invasion;
* with immunotherapy or radiotherapy contraindication;
* ever suffered with malignant tumor;
* having peripheral nervous system disorder or dysphrenia;
* with no legal capacity,medical or ethical reasons affecting research proceeding;
* participating other clinical trials simultaneously;
* adopting other anti-tumor medicine excluding this research;
* Patients with immunodeficiency, such as primary immunodeficiency syndrome or organ transplant recipients
* Human immunodeficiency virus (HIV)-positive patients
* the researchers considering it inappropriate to participate in the study.
* Patients with immune system diseases

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | From date of randomization until the date tumor volume has reduced, assessed up to 36 months
  The proportion of patients whose tumor volume has reduced to a predetermined value and can maintain the minimum time limit is the sum of complete and partial mitigation.
Progression-free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The time between the start of randomization and the progression of the tumor (any aspect) or (for any reason) death
Overall Survival | From date of randomization until date of death from any cause, assessed up to 36 months
  Time from randomization to death for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department of The First Affilliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No